CLINICAL TRIAL: NCT01934348
Title: Psychological First Aid for Victims of Crime
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH091203 (NIH)
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2013-08

CONDITIONS: Posttraumatic Stress Disorder; Depression; Substance Use
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders | interventions — Psychological First Aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological First Aid (Experimental): Behavioral intervention delivered to crime victims during 2-3 in-person interactions within 1 month of the assault.
  Interventions: Behavioral: Psychological First Aid
- Usual victim advocacy services (Active Comparator): Standard victim advocacy services delivered to crime victims within 1 month of the assault.
  Interventions: Behavioral: Usual victim advocacy Services

INTERVENTIONS:
Behavioral: Psychological First Aid
  Arms: Psychological First Aid
Behavioral: Usual victim advocacy Services
  Arms: Usual victim advocacy services

SUMMARY:
This study aims to implement and refine research protocols required for a full-scale randomized controlled trial of Psychological First Aid (PFA) for adult victims of crime. PFA is a promising acute intervention designed to reduce the severity and duration of trauma-related distress. Law Enforcement Victim Advocates are being trained to implement PFA with adult crime victims. A pilot trial is comparing PFA to usual victim advocacy services on key psychiatric outcomes from baseline through 4 months post-baseline.

DETAILED DESCRIPTION:
Criminal victimization represents a major public health problem in the United States. As many as one-third of adults have been the victim of a violent crime (rape/sexual assault, physical assault, or armed robbery) during their lifetime, and individuals exposed to violence are at risk for developing chronic psychiatric problems, including posttraumatic stress disorder (PTSD), depression, and substance abuse.

The high prevalence of psychopathology among crime victims underscores the importance of effective interventions for this population. As such, considerable work has validated formal treatments for victims who have already developed chronic trauma-related difficulties. Very little effort, however, has been devoted to testing acute interventions that can be implemented soon after a crime event (i.e., within 4 weeks) with the ultimate aim of preventing longer-term psychiatric problems.

Despite the limited research on acute interventions for crime victims, researchers recently developed an acute intervention called Psychological First Aid (PFA) for individuals exposed to natural disasters or other catastrophic events. Important for present purposes, however, researchers have argued that the primary PFA components (Contact and Engagement, Stabilization, Information Gathering, Safety Planning, Practical Assistance, Connection with Social Supports, Information on Coping, and Linkage with Collaborative Services) also have direct relevance for victims of crime. Thus, we propose that PFA could represent an ideal approach for responding to the acute needs of crime victims, with the goal of reducing their risk for development of chronic psychiatric problems. Importantly, although PFA has been strongly advocated by trauma experts, there have been no empirical tests of the model, highlighting the importance of the proposed research.

Thus, this R34 project aims to implement and refine research protocols required for a full-scale randomized controlled trial of PFA for crime victims. Specifically, this project will examine the feasibility of a protocol for recruiting, assessing, and retaining acute crime victims in the study (Aim 1). Additional preliminary work that is essential for treatment research also will be completed, including the development and evaluation of a PFA fidelity instrument (Aim 2) and the refinement and testing of protocols for training paraprofessionals (i.e., Victim Advocates) to deliver PFA with a high level of fidelity (Aim 3). Finally, a controlled pilot study will examine the effects of PFA on the key psychiatric outcomes (Aim 4).

ELIGIBILITY:
Inclusion Criteria:

* Victim of a rape/sexual assault, physical assault, or armed robbery
* Experience of a physical injury or perceived life threat during the assault

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in the frequency and severity of posttraumatic stress disorder symptoms as measured by the National Stressful Events PTSD Scale | Baseline, 1-, 2-, & 4-months post-baseline
Change in the frequency and severity of general anxiety, depression, and somatic symptoms as measured by the Brief Symptom Inventory-18 | Baseline, 1-, 2-, & 4-months post-baseline
Change in the frequency and severity of substance use as measured by the Addiction Severity Index-Self Report | Baseline, 1-, 2-, & 4-months post-baseline

SECONDARY OUTCOMES:
Change in the frequency of exposure to traumatic events as measured by the Trauma Assessment for Adults-Brief Version | Baseline, 1-, 2-, & 4-months post-baseline
Change in the level of adaptive functioning as measured by the Social Adjustment Scale-Self Report | 1-, 2-, & 4-months post-baseline
Change in the utilization of formal treatment services as measured by the Service Utilization Form | 1-, 2-, & 4-months post-baseline
Change in the frequency of contact between Victim Advocates and crime victims as measured by the Advocate Contact Form | Up to 9 months following randomization of the advocates to the PFA and usual services conditions
Change in the level of PFA implementation by Victim Advocates as measured by the PFA Fidelity Form | Up to 9 months following randomization of the advocates to the PFA and usual services conditions

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. McCart, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Charleston County Sheriff's Office, Charleston, South Carolina
  - City of Charleston Police Department, Charleston, South Carolina